CLINICAL TRIAL: NCT01471184
Title: A Double-Blind, Randomized, Cross-Over Study of The Effects of Ectoin® Allergy Nasal Spray and Ectoin® Allergy Eye Drops Compared to Placebo, in Patients With Allergic Rhinitis and Allergic Conjunctivitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: The Effects of Ectoin® Allergy Nasal Spray and Ectoin® Allergy Eye Drops Compared to Placebo
Acronym: PPL-003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P2JH09001
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis
Keywords: Allergic Rhinitis; Conjunctivitis; Bitop; Eye; Eye Drops; Nasal Spray; Total Nasal Symptom Score; Total Ocular Symptom Score; AUC
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ectoin® Eye Drops/Nasal Spray (Experimental): Eye Drops/Nasal Spray
  Interventions: Device: Ectoin® Allergy Nasal Spray and Ectoin® Allergy Eye Drops
- Placebo Eye Drops/Nasal Spray (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Ectoin® Allergy Nasal Spray and Ectoin® Allergy Eye Drops
  Arms: Ectoin® Eye Drops/Nasal Spray
Device: Placebo — Placebo Eye Drops/Nasal Spray
  Arms: Placebo Eye Drops/Nasal Spray

SUMMARY:
The primary objective of this study is to assess the relative efficacy of Ectoin® Allergy Eye Drops and Ectoine® Allergy Nasal Spray compared to placebo, by evaluating Total Nasal Symptom Score (TNSS) and Total Ocular Symptom Score (TOSS).

The secondary objectives are :

* To evaluate the relative efficacy of Ectoin® Allergy Eye Drops and Ectoin® Allergy Nasal Spray compared to placebo by evaluating Total Non Nasal Symptom Score (TNNSS), congestion symptom scores, red eye symptom scores, watery eye symptom scores, itchy eye symptom scores, and by evaluating the mean cross-sectional area (MCA) using acoustic rhinometry (AcR).
* To assess the change from baseline (post-EEC from pre-EEC) in inflammatory parameters of nasal secretions, comparing Ectoin® Allergy Eye Drops and Ectoin® Allergy Nasal Spray to placebo at each post-treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a clinical history of SAR with seasonal onset and offset of nasal and ocular allergy symptoms at least during each of the last two ragweed allergy seasons.
2. Adults (males and females) aged 18 to 65, inclusive.
3. Patients must have documentation of a positive skin test within 12 months of screening to ragweed or a positive skin prick and/or intradermal test for ragweed allergen at Visit 1. A positive response is defined as a wheal diameter of at least 3 mm larger than the negative control for the skin prick test or at least 7 mm larger than the negative control for the intradermal test.
4. Non-pregnant, non-lactating women not of childbearing potential who are post-menopausal [defined as at least 6 months natural spontaneous amenorrhea], or are surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Surgical sterility should be supported with clinical documentation.

   Females must have a confirmed absence of pregnancy according to a negative serum pregnancy test or urine pregnancy test at the times described in Section 11.

   Female subjects of child bearing potential must agree to use a reliable and highly effective method of birth control with a low failure rate (i.e. less than 1% per year) when used consistently and correctly (e.g. implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partners) during the trial, as judged by the investigator. For subjects using a hormonal contraceptive method, information regarding the product under evaluation and its potential effect on the contraceptive should be addressed.
5. In generally good health on the basis of medical history and physical examination.
6. Willingness to attend all study visits.
7. Capable of following and understanding instructions.
8. Willing and able to provide written informed consent prior to initiation of any study procedures, including initiation of washout of any concomitant medications.

Exclusion Criteria:

1. Asthma based on medical history or investigator judgment (stable mild asthmatics may be included).
2. Current smoker and ex-smokers with more than 10 pack years smoking history. One pack year is defined as 20 cigarettes/day for 1 year. Smoking must have been stopped more than 6 months ago
3. History of lower or upper airway infection in the last four weeks prior to screening.
4. Clinically significant physical findings of nasal anatomical deformities causing greater than 50% obstruction based on the clinical estimate of the investigator, including nasal polyps, septal defects or other clinically significant respiratory tract malformations, nasal piercing, recent nasal biopsy, nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa within 60 days prior to the Screening Visit.
5. Pregnancy or breastfeeding, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period, or for 30 days following the study period.
6. Currently participating in a clinical trial or has been exposed to an investigational treatment within the 30 days prior to the Screening Visit.
7. A known or suspected hypersensitivity, and/or contraindication to any of the ingredients of the investigational products.
8. History of alcohol or drug abuse, as judged by the investigator, within the two years prior to the Screening Visit.
9. Use of any of the prohibited medications within the identified exclusion periods (see Section 3.2.4)
10. Any acute or chronic disease that, in the opinion of the investigator, would affect the study objectives or subject safety (e.g., Diabetes mellitus type I, malignant neoplasia, chronic renal failure, inflammatory diseases of liver or kidneys, emphysema, bronchiectasis).
11. Any clinically significant (as determined by the investigator) psychiatric and/or psychological disorders, including impairment of cooperation (e.g. alcohol or drug abuse).
12. Patients not able to follow study procedures (e.g. language problems, psychological disorders).
13. Suspected non-compliance to study protocol. Non-compliance is e.g. application of less than 60% (according to post treatment container's weight) or missing more than one application on either of the last two days before EEC.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Ectoin Allergy Eye Drops and Ectoine Allergy Nasal Spray assess the relative efficacy | From baseline to end of treatment at 13 days
  The primary objective of this study is to assess the relative efficacy of Ectoin® Allergy Eye Drops and Ectoine® Allergy Nasal Spray compared to placebo, by evaluating Total Nasal Symptom Score (TNSS) and Total Ocular Symptom Score (TOSS).

SECONDARY OUTCOMES:
Relative efficacy of Ectoin Allergy Eye Drops and Ectoin Allergy Nasal Spray compared to placebo | From baseline to end of treatment at 13 days
  To evaluate the relative efficacy of Ectoin® Allergy Eye Drops and Ectoin® Allergy Nasal Spray compared to placebo by evaluating Total Non Nasal Symptom Score (TNNSS), congestion symptom scores, red eye symptom scores, watery eye symptom scores, itchy eye symptom scores, and by evaluating the mean cross-sectional area (MCA) using acoustic rhinometry (AcR).

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada